CLINICAL TRIAL: NCT00609219
Title: Administration of EBV-Specific T-Lymphocytes to Patients With EBV-Positive Nasopharyngeal Carcinoma
Brief Title: T-Lymphocytes in Treating Patients With Epstein-Barr Virus-Positive Nasopharyngeal Cancer, NPC
Acronym: NPC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Helen Heslop, Professor, Director-Adult Stem Cell Transplant Program, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-9935-NPC; NPC; NCT00074594 (obsolete NCT alias)
Record Dates: First submitted 2008-02-02; First posted 2008-02-06 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Head and Neck Cancer
Keywords: recurrent nasopharyngeal cancer; stage II nasopharyngeal cancer; stage III nasopharyngeal cancer; stage IV nasopharyngeal cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Nasopharyngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EBV specific CTL (Experimental): autologous EBV specific CTLs
  Interventions: Biological: autologous EBV specific CTLs

INTERVENTIONS:
Biological: autologous EBV specific CTLs — 30-40cc of peripheral blood will be used to generate EBV specific CTLs
  Group One:
  Day 0 - 2 x 10^7 cells/m2 Day 14 - 2 x 10^7 cells/m2
  Group Two:
  Day 0 - 2 x 10^7 cells/m2 Day 14 - 1 x 10^8 cells/m2
  Group Three:
  Day 0 - 1 x 10^8 cells/m2 Day 14 - 2 x 10^8 cells/m2
  Other Names: EBV specific CTLs

SUMMARY:
Patients have a type of cancer called nasopharyngeal cancer. This cancer has come back or not gone away or is at high risk for coming back after treatment (including the best treatment we know for nasopharyngeal cancer). We are asking patients to volunteer to be in a research study using special immune system cells called EBV-specific cytotoxic T lymphocytes, a new experimental therapy.

Most patients with nasopharyngeal cancer show evidence of infection with the virus that causes infectious mononucleosis, Epstein Barr virus (EBV), before or at the time of their diagnosis of nasopharyngeal cancer. EBV is found in the cancer cells of most patients with nasopharyngeal cancer, suggesting that it may play a role in causing this cancer. The cancer cells infected by EBV are able to hide from the body's immune system and escape destruction. We want to see if special white blood cells (called T cells) that have been trained to kill EBV-infected cells can survive in the patient's blood and affect the tumor.

We have treated other patients with different EBV positive cancers and have had variable results. Some patients have had some response to the treatment. Some patients have been cured by the treatment. It is not possible for us to predict if this treatment will work for nasopharyngeal cancer.

The purposes of this study are to find the largest safe dose of EBV specific cytotoxic T cells, to learn what the side effects are, and to see whether this therapy might help patients with nasopharyngeal cancer.

DETAILED DESCRIPTION:
We will first test a biopsy of the tumor (that has already been done) to see if your tumor cells are EBV positive. If the patient is eligible, we will then take 60-70 ml (12-14 teaspoons) of blood from them. We will use this blood to grow more of the T cells in the laboratory. We will first grow an EBV-infected cell line by infecting the blood with EBV virus. This line will then be irradiated so it cannot grow and used to stimulate the T cells. This stimulation will train the T cells to kill cells with EBV on their surface. We will then grow these EBV-specific CTLs by more stimulation with EBV infected cells and a growth factor called Interleukin 2. Next, we will test the T cells to make sure that they kill the EBV-infected cells. If the number of T cells produced is low, we may need to obtain additional blood samples to make these cells.

The cells (which are the patient's own T cells) will be injected into them over 10 minutes, after pretreatment with Tylenol and Benadryl. A total of two doses will be given two weeks apart. All of the Treatments will be given by the Center for Cell and Gene Therapy at Texas Children's Hospital or the Methodist Hospital.

We will follow the patient in the clinic after the injections. To learn more about the way the T cells are working and how long they last in the body, an extra 10-60 mls (2-12 teaspoons) of blood will be taken before the infusion and 3-4 days after the infusion (this is optional). Up to 40 ml (8 teaspoons) of blood will also be drawn at 1, 2, 4 and 6 weeks post-infusion, and then at 3, 6, 9, and 12 months. The blood may be drawn from the patient's central line at the time of the regular blood tests. We will use this blood to look at the immune response to the patient's cancer. Over the course of the study, up to 29 tablespoons of blood will be drawn.

Patients will also have repeat scans at 8 weeks after the first injections. If these show stable or improving disease they may (if the patient wishs) receive up to 6 extra doses of cells. These would be given every 1-3 months. If the patient has additional injections of cells after the first two infusions, we will take extra blood tests before each infusion, at the end of each infusion, 3-4 days after each infusion (day optional depending on patient preference), and at 1 and 2 weeks after each infusion. We will also do an extra scan between 1 and 3 months after the last infusion. Follow up will then continue every 3 months and will continue until 12 months after the last infusion.

ELIGIBILITY:
Inclusion Criteria:

* All patients with NPC in first or subsequent relapse or with primary refractory disease or high risk (T3 or T4, or node positive disease) in whom the EBV genome or antigens have been demonstrated in tissue biopsies will be eligible for this trial. -Patients with a life expectancy >6 weeks
* Patients with a Karnofsky score of >/= 50
* No severe intercurrent infection.
* Patient, parent/guardian able to give informed consent.
* Patients with bilirubin <2x normal, SGOT <3x normal, and Hgb >8.0
* Patients with a creatinine <2x normal for age
* Patients should have been off other investigational therapy for one month prior to entry in this study.

Exclusion Criteria:

-Patients with a life expectancy of <6 weeks. -Patients with a Karnofsky score of < 50. -Patients with a severe intercurrent infection. -Patient, parent/guardian unable to give informed consent. -Patients with a bilirubin >2x normal. SGOT >3x normal or abnormal prothrombin time. -Patients with a creatinine >2x normal for age -Due to unknown effects of this therapy on a fetus, pregnant women are excluded from this research. The male partner should use a condom.

Note: Patients who would be excluded from the protocol strictly for laboratory abnormalities can be included at the investigators discretion after approval by the CAGT Protocol Review Committee and the FDA reviewer.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2001-08; Primary Completion 2007-10 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Safety of two IV injections of autologously derived Epstein-Barr virus (EBV)-specific cytotoxic T-lymphocytes (CTLs) | 6 weeks
  Patients will be enrolled at the first dose level and followed for six weeks after the second dose (which will constitute a course) for evaluation of any critical toxicity

SECONDARY OUTCOMES:
the survival, immunological efficacy and anti-tumor effects of EBV specific cytotoxic T-lymphocyte lines. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Helen E. Heslop, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Texas Children's Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas

REFERENCES:
- [Background] Louis CU, Straathof K, Bollard CM, Ennamuri S, Gerken C, Lopez TT, Huls MH, Sheehan A, Wu MF, Liu H, Gee A, Brenner MK, Rooney CM, Heslop HE, Gottschalk S. Adoptive transfer of EBV-specific T cells results in sustained clinical responses in patients with locoregional nasopharyngeal carcinoma. J Immunother. 2010 Nov-Dec;33(9):983-90. doi: 10.1097/CJI.0b013e3181f3cbf4. PMID 20948438
- [Result] Straathof KC, Bollard CM, Popat U, Huls MH, Lopez T, Morriss MC, Gresik MV, Gee AP, Russell HV, Brenner MK, Rooney CM, Heslop HE. Treatment of nasopharyngeal carcinoma with Epstein-Barr virus--specific T lymphocytes. Blood. 2005 Mar 1;105(5):1898-904. doi: 10.1182/blood-2004-07-2975. Epub 2004 Nov 12. PMID 15542583